CLINICAL TRIAL: NCT00606112
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled Ascending IV Single-Dose Tolerance and Pharmacokinetic Study of Trodusquemine (MSI-1436) in Obese Type 2 Diabetics
Brief Title: A Single Dose, Tolerance and Pharmacokinetic Study in Obese or Overweight Type 2 Diabetic Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Responsible Party: Michael Gast, MD, PhD, Genaera Corporation
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSI-1436C-103
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — 3-N-1(spermine)-7, 24-dihydroxy-5-cholestane 24-sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Trodusquemine (MSI-1436)
- 2 (Placebo Comparator)
  Interventions: Drug: Trodusquemine (MSI-1436)
- 3 (Placebo Comparator)
  Interventions: Drug: Trodusquemine (MSI-1436)
- 4 (Placebo Comparator)
  Interventions: Drug: Trodusquemine (MSI-1436)

INTERVENTIONS:
Drug: Trodusquemine (MSI-1436) — A single dose will be administered on Day 0. Doses are 3mg/m2 in cohort 1, 6mg/m2 in cohort 2, 10mg/m2 in cohort 3 and 15mg/m2 in cohort 4/

SUMMARY:
The purpose of this study is to evaluate the safety and tolerance of a single intravenous (through a vein) dose of trodusquemine (MSI-1436) in obese, type 2 diabetics.

Different amounts of trodusquemine (MSI-1436) will be given to each volunteer group throughout the study.

Another purpose is to evaluate the pharmacokinetics (PK - the study of the way the drug enters and leaves the blood and tissues over time) of trodusquemine (MSI-1436).

Finally, this study will also determine whether trodusquemine (MSI-1436) has any effect on appetite, mood or behavior, and selective biomarkers (substances in your blood that may change in response to the study drug).

ELIGIBILITY:
Inclusion Criteria:

1. male or female obese or overweight type 2 diabetic subjects, between 18 and 55 years old (inclusive)
2. either treatment naive or who are inadequately controlled on either metformin alone or metformin in combination with a sulfonylurea. Subjects on metformin in combination with a sulfonylurea will be allowed a 2 week period to wash out the sulfonylurea before dosing.
3. have a fasting blood sugar of ≥ 100 mg/dL, hemoglobin A1C ≥ 7.5% (but ≤ 11.0%). Subjects on a combination of metformin and sulfonylurea must have a hemoglobin A1C ≥ 7.5% (but ≤ 10.0%);
4. non-smoker
5. body mass index (BMI) of 27-40 kg/m2

Exclusion Criteria:

1. likely allergy or sensitivity to any components of Trodusquemine (MSI-1436) for Injection based on known allergies to drugs of the same class;
2. any subject with a history of allergy (rash, hives, breathing difficulty, etc.) to any medications, either prescription or nonprescription, including dietary supplements or herbal medications;
3. any subject with a history of severe allergy or bronchial asthma;
4. a clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, gastrointestinal, cardiovascular (except hyperlipidemia or controlled hypertension), pulmonary (including chronic asthma), endocrine (except diabetes), central nervous, or hematologic systems, or recent clinically significant surgery;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance of a single intravenous dose of trodusquemine (MSI-1436) in obese, type 2 diabetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kipnes, MD, Principal Investigator — dgd Research; Gilbert R. Weiner, D.O. AOBFP, Principal Investigator — Allied Research International
Locations (1):
- dgd Research, San Antonio, Texas, United States